CLINICAL TRIAL: NCT00396734
Title: The Effects of Modafinil and Topiramate on Brain Mechanisms Underlying Cue-induced Cocaine Craving and Dependence in Methadone Maintained Cocaine Dependent Patients.
Brief Title: The Effects of Pharmacotherapy on Brain Mechanisms Underlying Cocaine Dependence.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant was not renewed
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr Arik Zukert, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 281006-HMO-CTIL
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Opioid-Related Disorders; Cocaine-Related Disorders
Keywords: Imaging; cocaine; methadone; craving; PET; FDG; D2; Modafinil; Topiramate
MeSH Terms: conditions — Opioid-Related Disorders; Cocaine-Related Disorders | interventions — Modafinil; Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Provigil (Modafinil) — Increase from 100mg to 400mg during 1 month of treatment
Drug: Topamax (Topiramate) — Increase from 25mg to 200mg in one month (double every week)

SUMMARY:
The overall aim of this project is to use an advanced brain imaging technique, PET, in order to monitor the progress of pharmacotherapy with modafinil or topiramate for cocaine dependence in methadone-maintained patients who use cocaine in addition. Comparisons will be made within the cocaine dependent methadone maintained subjects, between the start and end of treatment, and between the two medications. This is the first systematic research study of pharmacological treatment for cocaine dependence in Israel. This study is of major clinical use, with implications for the treatment of cocaine dependence in poly-drug abusers in Israel. Successful pharmacotherapy for cocaine dependence is expected in reduction in cue-induced subjective craving and in glucose metabolism in brain areas elicited by cocaine craving. Metabolic activity in regions that are activated by craving should be correlated with dopamine DRD2 receptor occupancy in all patients.

DETAILED DESCRIPTION:
SPECIFIC AIMS

1. To try to elucidate the brain mechanisms underlying cocaine dependence and craving in co-morbid cocaine-dependent patients. For this purpose we shall trigger craving for cocaine by exposure to a videotape showing cocaine use and then measure brain metabolic activity using Positron Emission Tomography (PET) and [18F] Fluorodeoxyglucose (FDG)
2. To evaluate dopamine binding in the brain in the early stage, and at the end of treatment. For this purpose the patients will undergo brain imaging of the dopamine receptor DRD2 by using PET with [11C] raclopride. This is a well established procedure for quantifying the effects of drugs such as amphetamine and cocaine on the brain.
3. To investigate the association between subjective measures of craving for cocaine and the level of dopamine DRD2 receptor occupancy in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Methadone-maintained cocaine-dependent patients use between 1g to 2g a day; 1 to 3 times a week

Exclusion Criteria:

* use more than 2g a day; 5 times a week to everyday
* Subjects who are diagnosed as suffering from psychotic illness according to DSM-IV (Axis 1)22, or with a history of CNS disease, a history of infection that might affect CNS (HIV, syphilis, cytomegalovirus, herpes), or a history of head injury with loss of consciousness,pregnant women.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Changes in cue-induced brain glucose metabolic activity (FDG) in PET after treatment. | 1 month
Changes in DRD2 receptor density measured by 11 C Raclopride in PET after treatment. | 1 month
Nr.of drug-free urine samples, time to first drug use, duration of longest abstinent period. | 1 month

SECONDARY OUTCOMES:
Craving and psychosocial functioning (e.g., employment status, criminal behavior). | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Aviv M Weinstein, Ph.D, Study Director — Hadassah Medical Organization; Roland Chisin, M.D, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel